CLINICAL TRIAL: NCT07023640
Title: Application of the CD73-Targeted Probe ⁶⁸Ga-DOTA-mPNE PET/CT Imaging in the Diagnosis of Malignant Tumors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCH-CD73-3
Record Dates: First submitted 2025-06-04; First posted 2025-06-17 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-06

CONDITIONS: Malignant Neoplasms of Brain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Malignant Neoplasms (Experimental)
  Interventions: Diagnostic Test: 68Ga-DOTA-mPNE

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTA-mPNE — PET/CT examination was performed after intravenous injection of 68GA-DOTA-mPNE tracer

SUMMARY:
This study aims to perform ⁶⁸Ga-DOTA-mPNE PET/CT imaging in patients with clinically suspected or confirmed malignant tumors, in order to evaluate tracer uptake in lesions and analyze CD73 expression levels. In a subgroup of up to 10 participants, dynamic PET/CT imaging will be conducted for up to 90 minutes post-injection to assess the tracer's biodistribution and pharmacokinetic properties.Correlation analyses with relevant clinical indicators (such as pathology, immunohistochemistry, and molecular markers) will be carried out to further assess the diagnostic performance and clinical value of ⁶⁸Ga-DOTA-mPNE PET/CT in guiding tumor diagnosis and treatment. This study is expected to provide a novel molecular imaging tool for malignancies and offer clear, intuitive PET/CT-based evidence to support clinical diagnosis, differential diagnosis, and therapeutic decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years, with an expected survival of ≥12 weeks.
2. No prior radiotherapy or chemotherapy; eligible for surgery or biopsy to obtain pathological diagnosis.
3. At least one measurable target lesion according to RECIST version 1.1 (Response Evaluation Criteria in Solid Tumors).
4. Written informed consent obtained and able to comply with follow-up requirements.

Exclusion Criteria:

1. Severe hepatic or renal dysfunction.
2. Women who are planning to conceive, currently pregnant, breastfeeding, or intend to have children during the study period are not eligible. Fertile participants must use effective contraception during the study.
3. Unable to lie flat for 30 minutes.
4. Refusal to participate in this clinical study.
5. Claustrophobia or other psychiatric disorders.
6. Any other condition deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-10 (Actual); Primary Completion 2026-06-17 (Estimated); Study Completion 2026-06-17 (Estimated)

PRIMARY OUTCOMES:
SUVmax | Time Frame: Day 1 (on the day of PET/CT imaging)
  The area of interest was delineated and the SUVmax value was measured by using the post-processing software built into the acquisition machine.

CONTACTS AND LOCATIONS:
Overall Officials: Xianzhong Zhang, PhD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China